CLINICAL TRIAL: NCT05888883
Title: Microbial Keratitis Sampling for Biomarker Discovery
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023/0017
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Microbial Keratitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be retained. Swab samples will undergo DNA extraction, amplification and sequencing for pathogens (bacterial and fungal) present within the sample. No human DNA will be studied.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Microbial Keratitis Participants: Up to 50 participants presenting with clinically suspected microbial keratitis will be recruited from the Princess Alexandra Eye Pavilion, NHS Lothian, Edinburgh
- Healthy Control Participants: Up to 20 participants with no history of microbial keratitis will be recruited.

SUMMARY:
The goal of this observational study is to identify prognostic and/or diagnostic signatures (biomarkers) related to microbial keratitis outcomes. We will compare tear and ocular swab samples from participants currently suffering from microbial keratitis to healthy control participants.

The primary study objective is to undertake analysis (proteomics and metabolomics) of microbial keratitis patient (and healthy control) ocular samples collected throughout the patient treatment course to better understand the ocular microenvironment and to identify candidate biomarkers for future targeted screening and validation studies.

The secondary study objective is to define the microorganisms in patients with microbial keratitis through a better understanding of the ocular surface micro/mycobiome (the resident bacteria and fungi) in health and disease

Participants will have their tears collected via capillary tube during their treatment course, and swabs of their conjunctiva collected at their first and final appointments.

DETAILED DESCRIPTION:
Microbial keratitis (MK) (infection of the cornea) is a leading cause of blindness globally with an incidence of >2m cases per year (particularly across Low and Middle Income Countries - LMICs), and a common acute eye disease in Edinburgh (~ 100 cases treated at the Princes Alexandra Eye Pavilion (PAEP) per year). MK is an "ophthalmic emergency" and even where gold-standard diagnostics and treatment are available, over 60% of MK patients are still left with visual impairment across LMICs, and >10% of patients require expensive and often unsuccessful surgical interventions such as corneal transplant. These permanent, debilitating outcomes are often attributed to an excessive and uncontrolled immune response, leading to scarring and corneal perforation.

Despite this, current diagnostic and treatment strategy targets only the invading pathogen and does not address the host response. Even where microbiological evaluation is conducted, the average culture-positive rate is just 50% and Gram-stain positivity is reported between 27.3%-61.6%2. Where microbiological evaluation is not possible, antimicrobials are prescribed empirically and often inappropriately, potentially contributing to the emergence of antimicrobial resistance (AMR) and worsening outcomes.

We are seeking to better understand the inflammatory response and the host-pathogen interactions to develop improved diagnostics and alternative treatment strategies. We propose to achieve this by studying the tears and the conjunctiva of those currently with, and without MK to identify biomarkers which can be utilised to achieve these goals.

Research Question: Can prognostic and diagnostic signatures (biomarkers) for MK be identified from patient ocular samples (tears and swabs)?

Hypothesis: Biomarkers will be identified through proteomic/metabolomic and micro/mycobiome analysis of patient ocular samples and these can provide us with more information about the disease and could inform the development of novel diagnostic platforms and possible alternative treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* 16 years old or older.
* Able to provide informed consent for themselves.
* Patient group: Appearances typical of a new infective keratitis of the cornea, in one eye only.
* Control group: healthy volunteers with no recent history (within 1 year) of MK or inflammatory eye condition.

Exclusion Criteria:

* <16 years old.
* Not able to provide consent for themselves.
* Patients with suspected viral rather than bacterial/fungal corneal infection, such as herpetic keratitis.
* Patients who present with MK in both eyes.
* Control group: Individuals receiving topical steroid or antimicrobial therapy to the eye, or any other form of systemic immunosuppression/antimicrobial drug.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with suspected microbial keratitis will be recruited and consented at their first presentation at the Ophthalmology Acute Referral Clinic, or on-call service at the Princess Alexandra Eye Pavilion, Edinburgh, UK.
  Healthy control volunteer participants will be recruited from the University of Edinburgh by email invitation or by word-of-mouth
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Globally measure, list and compare the peptides extracted from ocular tear samples of participants with and without the disease (microbial keratitis) throughout the infection course. | 5 years
  Identify any proteomic signatures of disease prognosis
Globally measure, list and compare the metabolites extracted from ocular tear samples of participants with and without the disease (microbial keratitis) throughout the infection course. | 5 years
  Identify any metabolomic signatures of disease prognosis

SECONDARY OUTCOMES:
Measure, list and compare microorganisms (bacteria and fungi) extracted from ocular swab samples of participants with and without the disease (microbial keratitis) | 5 years
  Relative abundance of bacterial/fungal species between groups

CONTACTS AND LOCATIONS:
Overall Officials: Naing Latt Tint, FRCOphth, Principal Investigator — NHS Lothian
Locations (1):
- Princess Alexandra Eye Pavilion (NHS Lothian), Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided